CLINICAL TRIAL: NCT03212092
Title: Reducing Aggressive Behaviour Among People With an Intellectual Disability Through Supplementation of Vitamins, Minerals and n-3 Fatty Acids
Brief Title: Reducing Aggression Among People With an Intellectual Disability
Acronym: PSYVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Erik J. Giltay, MD, PhD, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL60839.058.17
Record Dates: First submitted 2017-06-16; First posted 2017-07-11 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Aggression; Intellectual Disability
Keywords: Aggression; aggressive behavior; nutritional supplements; dietary supplements; vitamin, mineral; omega-3; n-3 fatty acids; intellectual disability
MeSH Terms: conditions — Aggression; Intellectual Disability; Calcinosis | interventions — Geritol; Minerals

STUDY DESIGN:
Intervention Model Description: The study is a pragmatic multicenter randomized double-blind placebo-controlled intervention trial with an intervention period of 4 months. Since the washout period of several components of dietary supplements is unknown we chose a parallel design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo with the appearance as the dietary supplements
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multivitamin, mineral & n-3 FA (Experimental): The daily supplementation of multivitamin- and mineral in 2 capsules and n-3 fatty acids in 2 softgel capsules.
  Interventions: Dietary Supplement: Multivitamin, mineral & n-3 FA
- Placebo (Placebo Comparator): The placebo consists of daily supplementation of 2 capsules with rice bran extract, hypromellose and 1.6 mg riboflavin. And 2 softgel capsules with a vegetable oil.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multivitamin, mineral & n-3 FA — The 2 multi vitamin capsules with the two multi vitamin softgel capsules will be handed out once a day during a meal by the staff of the care organization. The compliance will be registered
  Arms: Multivitamin, mineral & n-3 FA
Dietary Supplement: Placebo — The placebo of the multi vitamin capsules and the two multi vitamin softgel capsules will be handed out once a day during a meal by the staff of the care organization. The compliance will be registered
  Arms: Placebo

SUMMARY:
The study is an randomised controlled trial (RCT) to test whether supplementation of vitamins, minerals and n-3 fatty acids may reduce aggressive behavior in people with intellectual disabilities.

DETAILED DESCRIPTION:
Rationale: The prevalence of aggression among people with an intellectual disability is high. Previous studies have demonstrated the potential of multivitamin-, mineral-, and n-3 fatty acids (n-3FA) supplementation to reduce antisocial behavior and aggression among schoolchildren and prisoners.

Objective: To test the hypothesis that multivitamin-, mineral-, and n-3 FA supplementation reduces aggression among adolescents and young adults with an intellectual disability.

Study design: Pragmatic, randomised, double blind, placebo controlled, multicentre intervention study.

Study population: People with an intellectual disability aged between 12-39 years, living at a care or treatment facility or having day care, who have shown aggressive behaviour.

Intervention: During 16 weeks, people in the active condition receive 4 supplements daily: 2 Bonusan Multi Vital Forte Actief (Multi vitamin and mineral) and 2 Bonusan Omega-3 Forte (n-3 fatty acids) while people in the placebo condition receive 4 placebo capsules.

Main study parameters/endpoints: The main study parameter is the number of aggressive incidents from baseline to endpoint (16 weeks post baseline), as measured using the Dutch version of the Modified Overt Aggression Scale (MOAS).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Clients who wish to participate enter a 2-week run-in phase during which they take 4 placebo capsules daily. After positive evaluation of this phase clients are randomised to either the active or control condition. Participants will then start the daily use of 4 supplement capsules or 4 placebo capsules, which continues for 16 weeks. At baseline and endpoint 2 questionnaires will be administered: the Intellectual Disability Quality of Life (IDQOL-16) and the Dutch Healthy Diet Food Frequency Questionnaire (DHD-FFQ). Small hair and faeces samples will be collected at baseline and 16 weeks. The data collection will take less than an hour per client and will take place at the location where the client resides. Aggression incidents will be registered by staff members using the MOAS. Also a staff member will fill in the Social Dysfunction Aggression Scale (SDAS) at baseline and endpoint, measuring observed levels of aggression and social dysfunction. The risks of participating in this study are minimal. The use of the Bonusan Multi Vital Forte Actief, or similar supplements has not been associated with any significant health risks and side effects. Potential benefits of participating in this study is an increase in quality of life through improved nutritional status, as well as a reduction of aggressive incidents. As this is a pragmatic trial in which the main objective is to determine whether the use of supplements has the potential to reduce the number of aggressive incidents among adolescents and young adults with an intellectual disability, it is imperative to include these subjects.

ELIGIBILITY:
Inclusion Criteria:

* intellectual disability
* living or day care in a health care organization
* age 12 till 39 years
* has a at least once a week an aggressive incident.

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* people with Williams syndrome, hyperparathyroid or hemochromatosis.
* Current use of nutritional supplements and refusal to quit this use for the duration of the study.
* Failure to complete the two-week run-in phase.
* The use of the following medication: levothyroxine, methyldopa en levodopa

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Aggression | The aggression will be reported daily by the staff during a period of 18 weeks
  The amount of aggressive behavior registered with the Modified Overt Aggression Scale (MOAS).This is a four item aggression scale which distinguishes verbal aggression, aggression to objects, self-aggression and physical aggression to others.

SECONDARY OUTCOMES:
Aggression and anti-social behavior | At baseline and in the 18th week
  Aggressive- and anti-social behavior measured with the SDAS-11. An eleven item aggression scale. The severity of each item can range from 1 to 5 on a Likert scale.
Quality of Life IDQOL-16 | At baseline and in the 18th week
  Quality of life measured with the IDQOL-16.
Cortisol status | At baseline and in the 18th week
  The cortisol status measured with hair analyses.
Microbiome | At baseline and in the 18th week
  The micobiome measured with feces analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Giltay, MD, PHD, Principal Investigator — Leiden University Medical Center
Locations (7):
- Netherlands (7):
  - Trajectum, Zwolle, Overijssel
  - Gemiva-SVG, Gouda, South Holland
  - Schakenbosch, Leidschendam, South Holland
  - s Heeren Loo, Amersfoort
  - Amerpoort, Baarn
  - Syndion, Gorinchem
  - Amarant, Tilburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schoenthaler SJ, Bier ID. The effect of vitamin-mineral supplementation on juvenile delinquency among American schoolchildren: a randomized, double-blind placebo-controlled trial. J Altern Complement Med. 2000 Feb;6(1):7-17. doi: 10.1089/acm.2000.6.7. PMID 10706231
- [Background] Gesch CB, Hammond SM, Hampson SE, Eves A, Crowder MJ. Influence of supplementary vitamins, minerals and essential fatty acids on the antisocial behaviour of young adult prisoners. Randomised, placebo-controlled trial. Br J Psychiatry. 2002 Jul;181:22-8. doi: 10.1192/bjp.181.1.22. PMID 12091259
- [Background] Zaalberg A, Nijman H, Bulten E, Stroosma L, van der Staak C. Effects of nutritional supplements on aggression, rule-breaking, and psychopathology among young adult prisoners. Aggress Behav. 2010 Mar-Apr;36(2):117-26. doi: 10.1002/ab.20335. PMID 20014286
- [Background] Long SJ, Benton D. A double-blind trial of the effect of docosahexaenoic acid and vitamin and mineral supplementation on aggression, impulsivity, and stress. Hum Psychopharmacol. 2013 May;28(3):238-47. doi: 10.1002/hup.2313. Epub 2013 Apr 29. PMID 23625531
- [Background] Raine A, Cheney RA, Ho R, Portnoy J, Liu J, Soyfer L, Hibbeln J, Richmond TS. Nutritional supplementation to reduce child aggression: a randomized, stratified, single-blind, factorial trial. J Child Psychol Psychiatry. 2016 Sep;57(9):1038-46. doi: 10.1111/jcpp.12565. Epub 2016 May 11. PMID 27166583
- [Background] Tammam JD, Steinsaltz D, Bester DW, Semb-Andenaes T, Stein JF. A randomised double-blind placebo-controlled trial investigating the behavioural effects of vitamin, mineral and n-3 fatty acid supplementation in typically developing adolescent schoolchildren. Br J Nutr. 2016 Jan 28;115(2):361-73. doi: 10.1017/S0007114515004390. Epub 2015 Nov 17. PMID 26573368
- [Background] Gajos JM, Beaver KM. The effect of omega-3 fatty acids on aggression: A meta-analysis. Neurosci Biobehav Rev. 2016 Oct;69:147-58. doi: 10.1016/j.neubiorev.2016.07.017. Epub 2016 Jul 20. PMID 27450580
- [Derived] de Bles NJ, Gast DAA, van der Slot AJC, Didden R, van Hemert AM, Rius-Ottenheim N, Giltay EJ. Lessons learned from two clinical trials on nutritional supplements to reduce aggressive behaviour. J Eval Clin Pract. 2022 Aug;28(4):607-614. doi: 10.1111/jep.13653. Epub 2022 Jan 17. PMID 35040231